CLINICAL TRIAL: NCT04671394
Title: The Use of Diode Laser and Green Indocyanine Solution in Adjunct to Full-mouth Ultrasonic Debridement in the Treatment of Periodontitis: a Randomized Controlled Trial
Brief Title: Diode Laser and Green Indocyanine in the Non-surgical Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Luigi Guida, Full Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Laser/01
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients in the control group are treated by the same operator and received a sham laser treatment in which, after pocket irrigation with the photosensitizer solution, the laser tip is inserted in the pockets but the laser unit is kept off.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (FMUD + DLIG) (Experimental): Periodontal pockets are treated by ultrasonic debridement and, after 7 and 28 days, by irrigation with indocyanine green solution and diode laser irradiation.
  Interventions: Procedure: FMUD + DLIG
- Control (FMUD + ST) (Sham Comparator): Periodontal pockets are treated by ultrasonic debridement and, after 7 and 28 days, by sham therapy.
  Interventions: Procedure: FMUD + ST

INTERVENTIONS:
Procedure: FMUD + DLIG — Full-Mouth Ultrasonic Debridement + Diode Laser and Indocyanine Green solution
  Other Names: Diode laser: Fox ARC, Sweden & Martina, Due Carrare, Italy; indocyanine green photosensitizer solution: Emundo®, Sweden&Martina, Due Carrare, Padova, Italy
  Arms: Test (FMUD + DLIG)
Procedure: FMUD + ST — Full-Mouth Ultrasonic Debridement + Sham Treatment
  Arms: Control (FMUD + ST)

SUMMARY:
This is a parallel-group, randomized controlled clinical trial aimed to evaluate the clinical and microbiological effects of the adjunctive topical use of diode laser and green indocyanine in the full-mouth ultrasonic debridement of patients affected by periodontitis.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease affecting the supporting tissues of the teeth and is primarily caused by the subgingival inflammation induced by the bacterial oral biofilm. Several risk factors may condition its development and progression and, if untreated, periodontitis may lead to tooth loss and severe functional and aesthetic impairments.

A central role in the non-surgical treatment of periodontitis is played by the manual and ultrasonic debridement of supra and subgingival bacterial deposits. The benefit of a fully ultrasonic approach lies in the knowledge that removing radicular structure is not a prerequisite for periodontal healing.

However, non-surgical therapy has limitations due to limited access to some sites (furcation areas, concavities, grooves, distal sites of molars, and deep pockets), which may impair periodontal healing due to the persistence of pathogens and subsequent recolonization. In this context, the use of diode laser in combination with photoactivated solutions has been proposed as an adjunct treatment to conventional periodontal therapy to enhance the antibacterial effect and improve clinical effects, especially in areas of difficult access.

In view of theme relevance and the existence of conflicting results in the literature, the aim of the present parallel-group, randomized controlled clinical trial is to evaluate the clinical and microbiological effects of the adjunctive topical use of diode laser and indocyanine green (DLIG) in the full-mouth ultrasonic debridement (FMUD) of patients affected by periodontitis.

24 patients will be treated by FMUD and, after 7 days, randomly allocated half to the test and a half to the control group. In the test group, patients will receive an adjunctive treatment in periodontal sites with an initial pocket depth > 4mm consisting of the use of a diode laser device (Fox ARC, Sweden & Martina, Due Carrare, Italy) after pocket irrigation by a solution of indocyanine green (Emundo®, Sweden&Martina, Due Carrare, Padova, Italy), whereas the patients in the control group will receive sham treatment (ST). The same treatment will be repeated three weeks after in both the test and control groups.

Clinical assessment and microbiological analysis of subgingival plaque will be performed at baseline and after 3 and 6 months.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of moderate to severe periodontitis
* Systemic health

Exclusion criteria:

* Systemic diseases requiring antibiotic prophylaxis or other systemic medication that could affect the patient's clinical response
* Periodontal treatment within the last 12 months or systemic antibiotic intake in the last 3 months
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Probing depth (PD) reduction | 6 months
  The distance between the bottom of the pocket and the gingival margin recorded with a manual probe using a light force and measured to the closest millimeter

SECONDARY OUTCOMES:
Recession (REC) increase | 6 months
  The distance between the gingival margin and the cemento-enamel junction or the margin of the restoration.
Clinical Attachment Level (CAL) gain | Baseline, 3 and 6 months
  Calculated as PD plus REC.
Microbiological analysis | 6 months
  Semi-quantitative analysis by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Guida, Prof., Principal Investigator — University of Campania Luigi Vanvitelli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Annunziata M, Donnarumma G, Guida A, Nastri L, Persico G, Fusco A, Sanz-Sanchez I, Guida L. Clinical and microbiological efficacy of indocyanine green-based antimicrobial photodynamic therapy as an adjunct to non-surgical treatment of periodontitis: a randomized controlled clinical trial. Clin Oral Investig. 2023 May;27(5):2385-2394. doi: 10.1007/s00784-023-04875-w. Epub 2023 Jan 31. PMID 36719506